CLINICAL TRIAL: NCT02565719
Title: An Open-label, Randomized, Active Controlled, Parallel Comparison Study of the Safety and Efficacy of REP 2139-Mg in Combination With Pegasys® and Viread® and REP 2165-Mg in Combination With Pegasys® and Viread® in Patients With HBeAg Negative Chronic Hepatitis B
Brief Title: REP 2139-Mg and REP 2165-Mg Combination Therapy in Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REP 401
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- REP 2139-Mg with Viread and Pegasys (Experimental): REP 2139-Mg in combination with tenofovir disoproxil fumarate (Viread) and pegylated interferon alpha-2a (Pegasys).
  Interventions: Drug: REP 2139-Mg; Drug: Pegasys; Drug: Viread
- REP 2165-Mg with Viread and Pegasys (Experimental): REP 2165-Mg in combination with tenofovir disoproxil fumarate (Viread) and pegylated interferon alpha-2a (Pegasys).
  Interventions: Drug: Pegasys; Drug: Viread; Drug: REP 2165-Mg
- Viread and Pegasys with crossover to REP 2139-Mg and Pegasys (Active Comparator): Tenofovir disoproxil fumarate (Viread) and pegylated interferon alpha-2a (Pegasys) - crossover into add-on REP 2139-Mg therapy (triple combination) in patients with < 3 log reduction in serum HBsAg from baseline after 24 weeks of Pegasys exposure.
  Interventions: Drug: REP 2139-Mg; Drug: Pegasys; Drug: Viread
- Viread and Pegasys with crossover to REP 2165-Mg and Pegasys (Active Comparator): Tenofovir disoproxil fumarate (Viread) and pegylated interferon alpha-2a (Pegasys) - crossover into add-on REP 2165-Mg therapy (triple combination) in patients with < 3 log reduction in serum HBsAg from baseline after 24 weeks of Pegasys exposure.
  Interventions: Drug: Pegasys; Drug: Viread; Drug: REP 2165-Mg

INTERVENTIONS:
Drug: REP 2139-Mg — REP 2139-Mg = magnesium chelate complex of REP 2139
  Other Names: not availalble
  Arms: REP 2139-Mg with Viread and Pegasys; Viread and Pegasys with crossover to REP 2139-Mg and Pegasys
Drug: Pegasys — immunotherapy
  Other Names: pegylated interferon alpha-2a
Drug: Viread — HBV RT polymerase inhibitor
  Other Names: tenofovir disoproxil fumarate
Drug: REP 2165-Mg — REP 2165-Mg = magnesium chelate complex of REP 2165
  Other Names: unaivalable
  Arms: REP 2165-Mg with Viread and Pegasys; Viread and Pegasys with crossover to REP 2165-Mg and Pegasys

SUMMARY:
NAPs have been previously shown to clear serum hepatitis B virus surface antigen (HBsAg) both preclinically (in duck HBV infected ducks) and in human patients. REP 2139-Ca mediated HBsAg clearance acts synergistically with immunotherapeutic agent pegylated interferon-alpha 2a to restore host immunological control of HBV infection. REP 2165 is a version of REP 2139 which has been shown preclinically to retain antiviral activity with lower accumulation in the liver.

Both REP 2139 and REP 2165 used in this protocol are formulated as magnesium chelate complexes, which improve their administration tolerability. This open label, randomized and controlled study will examine the safety and efficacy of REP 2139-Mg and REP 2165-Mg therapy in patients with HBeAg negative chronic hepatitis B when used in combination with tenofovir disoproxil fumarate and pegylated interferon alpha-2a.

DETAILED DESCRIPTION:
Nucleic acid polymers (NAPs) utilize the sequence independent properties of phosphorothioated oligonucleotides to target apolipoprotein interactions involved in the formation of HBV subviral particles (SVPs) which are comprised mainly of the hepatitis B surface antigen protein (HBsAg). The effect of NAPs is to block the formation of SVPs inside infected hepatocytes which prevents their secretion. As SVPs account for > 99.99% of HBsAg in the blood, NAPs are an effective approach for clearing HBsAg from the serum of HBV infected patient.

Previous clinical trials have demonstrated that treatment with the NAP REP 2139 (REP 2139-Ca) results in the rapid and effective clearance ofHBsAg from the blood. This HBsAg removal has the immediate effect of unmasking the underlying, pre-existing anti-HBsAg (anti-HBs) response, allowing clearance of HBV virus from the blood.

Although REP 2139-Ca has been shown to be safe in human patients, it shares the same class effect as other phosphorothioate oligonucleotides in that it accumulates in the liver with repeated dosing. REP 2165 is a version of REP 2139 which is designed to have an increased rate of degradation to slow down liver accumulation while keeping its antiviral activity intact. The antiviral efficacy of REP 2165 has been shown to be comparable to REP 2139 in a pre-clinical model of HBV infection with significantly less accumulation in the liver. As such, REP 2165 is expected to have comparable antiviral efficacy in human patients with reduced liver accumulation during treatment.

HBsAg has important immunosuppressive effects in HBV infection which have been shown to block both adaptive and innate immune processes. Removal of HBsAg from the blood of patients removes this immunosuppressive effect.

Thus, an important additional effect of removal of HBsAg from the blood is to greatly enhance the effect of pegylated interferon alpha 2a. It is expected that elimination of serum HBsAg with REP 2139-Mg or REP 2165-Mg will lead to creation of a favourable immunological activation in the absence of HBsAg, appearance of free anti-HBs, clearance of HBV virions in the blood and synergistic immunostimulation with conventional dosing of pegylated interferon alpha-2a and improved control of HBV infection in the presence of tenofovir disoproxil fumarate (TDF). All patients will receive 24 weeks of monotherapy with TDF prior to entry into experimental or active comparator arms.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Males or females 18-55 years of age
3. HBsAg> 1000 IU / ml at screening
4. HBV DNA > 10000 copies / ml at screening
5. Seronegative for HIV, HCV, CMV (IgM) and HDV (anti-HDAg) as determined at screening visit
6. HBeAg negative, anti-HBe positive
7. Evidence of liver fibrosis at screening
8. Non cirrhotic: absence of advanced cirrhosis based on fibroscan evaluation at screening.
9. Willingness to utilize adequate contraception while being treated with REP 2139-Mg or REP 2165-Mg and for 6 months following the end of the treatment in the study

   * Any woman of childbearing potential (WOCBP) who agrees to use an effective methods of birth control for the entire duration of the study.
   * Sexually active men who agree to use an effective method of birth control if their partners are WOCBP for the entire duration of the study for 6 months following the end of treatment.
10. Body Mass Index (BMI) ≥ 18 kg/m2 and ≤ 30kg/m2 at screening (http://www.nhlbisupport.com/bmi/bmicalc.htm)
11. Adequate venous access allowing weekly intravenous therapies and blood tests

Exclusion Criteria:

1. Women with positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG).
2. Breast-feeding women.
3. HBeAg positive as determined at screening visit
4. Positive HCV antibody, or HIV-1/HIV-2 or CMV antibody (IgM) or anti-HDV antibody test at screening
5. Evidence of chronic liver disease caused by diseases other than chronic HBV infection (such as but not limited to: severe NAFLD, Wilson's disease, hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, significant biliary disease, nonalcoholic hepatic steatosis and toxin exposure).
6. Medical History and Concurrent Diseases

   1. Current evidence of or history of variceal hemorrhage, hepatic encephalopathy, or ascites requiring diuretics or paracentesis or evidence of any of these findings on physical examination performed at screening
   2. Documented or suspected HCC as evidenced by previously obtained imaging studies or liver biopsy.
   3. Current evidence of or history of pancreatitis
   4. Current evidence of or history of renal dialysis, including hemodialysis or peritoneal dialysis
   5. History of bone marrow or organ transplant (other than cornea or hair), including liver transplant, or therapy with an immunomodulatory agent, cytotoxic agent, or systemic corticosteroids within 2 months of screening
   6. Current or known history of cancer (except adequately treated in situ carcinoma of the cervix, or basal or squamous cell carcinoma of the skin) within 5 years prior to screening
   7. Subjects with clinically significant ECG abnormalities (indicative of arrhythmia, myocardial ischemia or other serious cardiovascular disorder) at the time of screening in the opinion of the investigator
   8. Active substance abuse, such as alcohol, or inhaled or injected drugs, as defined by Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV), Diagnostic Criteria for Drug and Alcohol Abuse (see Appendix 1) within 12 months prior to screening.
   9. The use of illicit drugs within the past two years prior to screening.
   10. Prior or current history of cardiomyopathy or significant ischemic cardiac or cerebrovascular disease, including history of angina, myocardial infarction, or interventional procedure for coronary artery disease (including angioplasty, stent procedure, or cardiac bypass surgery)
   11. Confirmed uncontrolled hypertension (patients with screening systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg should be excluded unless discussed with Replicor Inc.)
   12. Presence of diabetes (controlled or uncontrolled).
   13. Prior or current history of clinically significant hemoglobinopathy or hemolytic anemia
   14. History of or evidence of hyperthyroidism at screening.
   15. Subjects with pre-existing ophthalmologic disorders considered clinically significant on eye exam during physical examination.
   16. Prior or current history of severe chronic obstructive pulmonary disease, interstitial lung disease or sarcoidosis
   17. History of immunologically mediated disease (including but not limited to, rheumatoid arthritis, inflammatory bowel disease, moderate to severe psoriasis [mild psoriasis is allowed], and systemic lupus erythematosus)
   18. History of or current severe psychiatric disease, especially untreated or unstable depression, psychotic disorder such as bipolar disease and history of hospitalization for suicidal ideation/attempt
   19. Active seizure disorder as defined by either untreated seizure disorder or continued seizure activity within the past year prior to screening despite treatment with anti-seizure medication
   20. Has, in the opinion of the investigator, any physical exam findings, laboratory abnormalities, or other medical, social, or psychosocial factors that may negatively impact compliance or subject's safety by participation in this study; this should include conditions which may affect hematologic parameters such as prior or current history of porphyria cutanea tarda and/or hemophilia
   21. Fibroscan and Fibromax showing current evidence advanced cirrhosis at screening or known history of decompensated cirrhosis based on radiologic criteria or biopsy results and clinical criteria
   22. Poor venous access making IV infusion too difficult
   23. Inability to provide informed consent
   24. Inability or unwillingness to provide weekly blood samples.
   25. Patients not willing to come every week to receive therapy or to give blood.
7. Physical and Laboratory Test Findings

   1. Evidence of significant heavy metal load in whole blood as determined at pre-screening visit.
   2. Antinuclear antibody (ANA) titer ≥ 1:640, AMA or LKM-1antibody positive as determined at pre-screening visit
   3. Hemoglobin < 12.0 g/dL (males), < 10.0 g/dL (female) at screening
   4. Platelet count < 90,000/mm3as determined at screening visit
   5. Creatinine clearance (CrCl) (as estimated by Cockcroft and Gault) ≤50 mL/min or confirmed creatinine persistently>1.5 mg/dl as determined at screening visit
   6. Total serum bilirubin>25umol/L as determined at screening visit.
   7. INR ≥ 2.0 as determined at screening visit
   8. PTT ≥ 2.0 x ULN as determined at screening visit
   9. Serum albumin ≤ 3.5 g/dL (35 g/L) as determined at screening visit
   10. ALT >10x ULN as determined at screening visit
   11. ANC ≤ 1,500 cells/mm3 as determined at screening visit
   12. Diagnosed or suspected hepatocellular carcinoma as evidenced by screening alpha-fetoprotein (AFP) of ≥ 100 ng/mL. If AFP is ≥ 50 ng/mL and < 100 ng/mL, absence of mass/findings suspicious for HCC must be demonstrated by ultrasound/CT/MRI within the screening period.
   13. Diabetes mellitus as evidenced by HbA1C ≥ 8.5% at screening
   14. QTc interval > 500 msec.
8. Known hypersensitivity to drugs with a similar biochemical structure to REP 2139-Mg or REP 2165-Mg (e.g. other phosphorothioate oligonucleotides) or Pegasys® (e.g. other interferons), Zadaxin® or Viread® (e.g. other nucleoside analog polymerase inhibitors such as entecavir).
9. Any other criteria or known contraindication that would exclude the subject from receiving REP 2139-Mg, REP 2165-Mg, Pegasys® or Viread®.
10. Prisoners or subjects who are involuntarily incarcerated.
11. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
12. Employees, family members, or students of the investigator or clinical site
13. Individuals who participated in another clinical study of a medicinal product or medical device within 90 days of signing Informed Consent Form
14. Concomitant Treatments with any of the following medications:

    1. Heparin
    2. Coumadin
    3. Blood products within 30 days prior to study enrollment
    4. Hematologic growth factors within 90 days prior to study enrollment
    5. Use of any investigational product within 1 year prior to study enrollment
    6. Systemic antibiotics, antifungals, or antivirals for treatment of active infection within 14 days of enrollment.
    7. Previous exposure to immunotherapy with 6 months prior to enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 48 or 72 weeks (treatment duration) + 48 weeks (follow-up)
  Patients will be assessed weekly for adverse events including symptoms and laboratory abnormalities

SECONDARY OUTCOMES:
Number of patients with reduction of serum HBsAg | Every two weeks for 48 or 72 weeks (treatment duration) + 48 weeks (follow-up)
  The primary action of NAPs is to lower serum HBsAg. This effect is monitored throughout treatment and for 48 weeks following treatment.
Number of patients with controlled HBV infection following treatment | 48 weeks follow-up (after completion of 48 or 72 weeks of treatment)
  The synergistic antiviral effect of HBsAg removal and immunotherapy has restored immunological control of HBV mono-infection in human patients which has persisted after treatment was stopped. The persistence of immunological control of HBV infection observed in this study will be followed for 48 weeks after treatment has stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Pantea, M.D., Principal Investigator — Infectious Diseases Department, State University of Medicine and Pharmacy, Infectious Clinical Hospital (n.a. Toma Clorba), Chisinau, Moldova, Republic of 2004
Locations (3):
- Moldova (3):
  - Infectious Clinical Hospital (n.a. Toma Ciorba) Department 5, Chisinau
  - Infectious Clinical Hospital (n.a. Toma Ciorba), Department 4, Chisinau
  - Repiblican Clinical Hospital (ARENSIA unit), Chisinau

REFERENCES:
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers inhibit duck hepatitis B virus infection in vitro. Antimicrob Agents Chemother. 2013 Nov;57(11):5291-8. doi: 10.1128/AAC.01003-13. Epub 2013 Aug 12. PMID 23939902
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers prevent the establishment of duck hepatitis B virus infection in vivo. Antimicrob Agents Chemother. 2013 Nov;57(11):5299-306. doi: 10.1128/AAC.01005-13. Epub 2013 Aug 12. PMID 23939904
- [Derived] Bazinet M, Anderson M, Pantea V, Placinta G, Moscalu I, Cebotarescu V, Cojuhari L, Jimbei P, Iarovoi L, Smesnoi V, Musteata T, Jucov A, Dittmer U, Gersch J, Holzmayer V, Kuhns M, Cloherty G, Vaillant A. Analysis of HBsAg Immunocomplexes and cccDNA Activity During and Persisting After NAP-Based Therapy. Hepatol Commun. 2021 Nov;5(11):1873-1887. doi: 10.1002/hep4.1767. Epub 2021 Jul 10. PMID 34558823
- [Derived] Bazinet M, Pantea V, Placinta G, Moscalu I, Cebotarescu V, Cojuhari L, Jimbei P, Iarovoi L, Smesnoi V, Musteata T, Jucov A, Dittmer U, Krawczyk A, Vaillant A. Safety and Efficacy of 48 Weeks REP 2139 or REP 2165, Tenofovir Disoproxil, and Pegylated Interferon Alfa-2a in Patients With Chronic HBV Infection Naive to Nucleos(t)ide Therapy. Gastroenterology. 2020 Jun;158(8):2180-2194. doi: 10.1053/j.gastro.2020.02.058. Epub 2020 Mar 6. PMID 32147484